CLINICAL TRIAL: NCT06848998
Title: Exercise and Cognition Among Stroke Survivors
Acronym: EXERCISES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17/EE/0409
Record Dates: First submitted 2025-02-05; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Aerobic Exercise; Resistance Exercise
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aerobic exercise (Experimental)
  Interventions: Behavioral: aerobic exercise
- Resistance exercise (Active Comparator)
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: aerobic exercise — 40 minutes of aerobic exercise, twice per week for six weeks.
  Sessions comprised of the following: 10-minute warm-up, 40-minute conditioning period as a circuit, and 10-minute cool-down.
  Aerobic exercises (for example, recumbent cycling, stepping, arm crank) commenced at an intensity of 40-50% heart rate reserve (HRR) and increased incrementally by 10% as tolerated, up to a maximum of 70-80%. All sessions were individually tailored as far as possible to participants' needs, abilities, and preferences.
  Arms: Aerobic exercise
Behavioral: Resistance exercise — 4 x resistance exercises (3 sets of 6 repetitions), twice per week for six weeks.
  Strengthening exercises (for example, resistance band work) were prescribed at an intensity that corresponded to 11-12 and incrementally increased to a maximum of 14-15, as tolerated, on the Borg Ratings of Perceived Exertion (RPE) 6-20 Scale. All sessions were individually tailored as far as possible to participants' needs, abilities, and preferences.
  Arms: Resistance exercise

SUMMARY:
This study aimed to: (1) identify a suitable cardiopulmonary exercise testing protocol for people with moderate to severe movement impairments after stroke by investigating the safety and feasibility of delivering two methods of CPET modes: treadmill with body-weight support (TBWS) and cycle ergometry (CE); and (2) explore the safety and feasibility of a delivering a 6-week exercise-based intervention or people with moderate to severe movement impairments after stroke, with a view to improve cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* Have provided informed consent,
* Are aged >18 years,
* Are more than 6 months post-stroke,
* Score 2-3 on the Functional Ambulation Category
* Can follow 1-stage commands i.e. sufficient communication/orientation for interventions in the trial.

Exclusion Criteria:

* Attending any other community exercise class/gym/walking group/rehabilitation class,
* A previous diagnosis of dementia or any other significant cognitive decline,
* Any musculoskeletal or neurophysiological disorder preventing participation in exercise,
* Have uncontrolled hypertension, atrial fibrillation, heart failure or diabetes.
* Weigh over 250lbs/113kg (due to weight restrictions on body-weight support harness on treadmill),
* Meeting any absolute or relative contraindication to exercise from American College of Sports Medicine (ACSM)

Contraindications to Exercise 2014, see below:

Absolute contraindications to exercise:

* A recent significant change in the resting ECG suggesting significant ischaemia, recent myocardial infarction (within 2 days) or other acute cardiac event
* Unstable angina
* Uncontrolled cardiac dysrhythmias causing symptoms or hemodynamic compromise
* Symptomatic severe aortic stenosis
* Uncontrolled symptomatic heart failure
* Actuate pulmonary embolus or pulmonary infarction
* Acute myocarditis or pericarditis
* Suspected or know dissecting aneurysm
* Acute systematic infection, accompanied by fever, body aches or swollen lymph glands

Relative contraindications to exercise:

* Left main coronary stenosis
* Moderate stenotic valvular heart disease
* Electrolyte abnormalities e.g. hypokalaemia, hypo-magnesia
* Severe arterial hypertensions i.e. systolic BP of >200mmHg and/or diastolic BP of >110mmHg at rest
* Tachydysrthythmia or bradydsrhythmia
* Hypertrophic cardiomyopathy and other forms of outflow tract obstruction
* Neuromuscular, musculoskeletal or rheumatoid disorders that are exacerbated by exercise
* High-degree atrioventricular block
* Ventricular aneurysm
* Uncontrolled metabolic disease e.g. diabetes, thyrotoxosis or myxedemia Chronic infectious diseases e.g. mononucleosis, hepatitis, AIDs
* Mental or physical impairment leading to inability to exercise adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | At baseline, and at the end of the intervention at 8 weeks
  Cardiorespiratory fitness was measured by means of a cardiopulmonary exercise test (CPET). Participants were allocated to the order of CPET mode: (1) treadmill with body weight support (TBWS) at baseline, followed by cycle ergometer (CE) post-intervention; or (2) CE at baseline, followed by TBWS post-intervention.
  For the treadmill protocol, participants were suspended by an overhead harness so that they were still weight-bearing but were able to walk using a reciprocal gait pattern with both feet flat on the treadmill. The starting speed was 0.5km/hr and was increased by 0.5 km/hr every one minute, until test termination.
  For the cycle ergometer protocol, participants pedalled on an upright ergometer at approximately 50 to 60 revolutions per minute, which increased by five watts, every minute, until test termination.

SECONDARY OUTCOMES:
Cognitive function | At baseline, and at the end of the intervention at 8 weeks
  Cognition was measured using the Montreal Cognitive Assessment (MoCA). The minimum score is 0 (indicating severe cognitive impairment) and the maximum score is 30 (indicating normal cognitive function). Scores of lower than 26 may indicate varying levels of cognitive impairment.
Activities of daily living | At baseline, and at the end of the intervention at 8 weeks
  Activities of daily living (ADL) was measured using the Barthel Index. Each activity (e.g., feeding, bathing, grooming) is scored based on the level of assistance required. The total score ranges from 0 to 100, with higher scores indicating greater independence.
Stroke specific quality of life | At baseline, and at the end of the intervention at 8 weeks
  Quality of life (QoL) was measured using the Stroke Specific Quality of Life Questionnaire (SSQoL). Each domain (e.g., mood, personality, social roles) consists of items scored from 1 to 5. The total SS-QOL score ranges from 49 to 245, where higher scores suggest a better stroke-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- University of East Anglia, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the lead contact (AW) upon reasonable request. This includes access to the full protocol and anonymised participant-level dataset.